CLINICAL TRIAL: NCT00039169
Title: An Uncontrolled Phase II Multi-Center Trial Evaluating Anti-Tumor Efficacy and Safety of BAY 59-8862 in Patients With Advanced Renal Cell Cancer
Brief Title: BAY 59-8862 in Treating Patients With Advanced Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069359; THERADEX-100386; BAYER-100386
Record Dates: First submitted 2002-06-06; First posted 2003-07-08 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — IDN 5109

INTERVENTIONS:
Drug: ortataxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BAY 59-8862 in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall tumor response rate, including complete response (CR) and partial response (PR) rate, in patients with advanced renal cell cancer treated with BAY 59-8862.
* Determine the overall survival in patients treated with this drug.
* Determine the time to progression in patients treated with this drug.
* Determine the duration of response (CR and PR) in patients treated with this drug.
* Determine the qualitative and quantitative toxicity profile of this drug in this patient population.
* Determine the pharmacokinetic profile of this drug in selected patients.

OUTLINE: This is a multicenter study.

Patients receive BAY 59-8862 IV over 1 hour on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months thereafter or for up to 2 years.

PROJECTED ACCRUAL: A total of 20-140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced renal cell cancer

  * Unresectable, refractory, and/or metastatic
* At least 1 measurable lesion

  * A CNS lesion cannot be the sole target lesion
  * Lesions within a previously irradiated field are not considered measurable
* No metastatic brain or meningeal tumors unless the patient received prior definitive therapy more than 6 months ago, has had a negative imaging study within the past 4 weeks, and is clinically stable with respect to the tumor at study entry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 2.0 times ULN (5.0 times ULN if hepatic involvement)
* PT, INR, and PTT less than 1.5 times ULN
* No chronic hepatitis B or C

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No clinically evident congestive heart failure
* No serious cardiac arrhythmias
* No prior coronary artery disease or ischemia

Other:

* No prior hypersensitivity to taxane compounds that was not considered clinically manageable with premedication
* No other malignancy within the past 3 years except carcinoma in situ of the cervix, adequately treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis, or T1)
* No substance abuse or medical, psychological, or social conditions that would preclude study compliance
* No active clinically serious infections
* No other condition that is unstable or would preclude study participation
* No grade 2 or greater pre-existing peripheral neuropathy
* No history of seizure disorder

  * Prior seizures related to brain metastases allowed provided that the patient has been seizure-free for at least 2 months
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 months since prior bone marrow or peripheral blood stem cell transplantation
* No more than 2 prior immunotherapy regimens (interleukin-2 or interferon only)
* At least 4 weeks since prior immunotherapy
* At least 3 weeks since prior biologic response modifiers (e.g., filgrastim [G-CSF])
* More than 4 weeks since prior thalidomide or bevacizumab
* No prior anticancer vaccines
* No concurrent prophylactic G-CSF
* Concurrent G-CSF or other hematopoietic growth factors for acute toxicity (e.g., febrile neutropenia) allowed
* Concurrent chronic epoetin alfa allowed provided no dose adjustment occurred within 2 months before study

Chemotherapy:

* No prior systemic cytotoxic chemotherapy
* No prior oxaliplatin
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Patients with prior metastatic brain or meningeal tumors:

  * No concurrent acute or tapered steroid therapy
  * Concurrent chronic steroid therapy allowed provided the dose is stable for 1 month before and after screening radiographic studies
* No hormonal therapy for renal cell cancer

Radiotherapy:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to target lesion identified for this study unless progression within the radiation portal is documented
* Concurrent palliative radiotherapy allowed provided:

  * No progressive disease
  * No more than 10% of bone marrow is irradiated
  * Radiation field does not encompass a target lesion
* No other concurrent radiotherapy

Surgery:

* At least 4 weeks since prior surgery
* No prior organ allograft

Other:

* At least 4 weeks since prior investigational drugs
* No other concurrent investigational therapy or approved anticancer therapy
* No concurrent illicit drugs or other substances that would preclude study
* Concurrent therapeutic anticoagulants (e.g., warfarin or heparin) allowed provided there is no prior evidence of underlying abnormality with PT, INR, or PTT
* Concurrent nonconventional therapies (e.g., herbs or acupuncture) or vitamin/mineral supplements allowed provided that they do not interfere with study endpoints
* Concurrent bisphosphonates for prophylaxis or bone metastases allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Marius Moscovici, MD, Study Chair — Pharma-Clinical
Locations (13):
- United States (11):
  - Scripps Clinic, La Jolla, California
  - Medical Consultants, Muncie, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - 206 Research Associates, Greenbelt, Maryland
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Billings Oncology Associates, Billings, Montana
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta